CLINICAL TRIAL: NCT04601792
Title: A Series of N-of-1 Trials on Bronchiectasis Treated With Traditional Chinese Medicine Based on Bayesian Model
Brief Title: A Series of N-of-1 Trials of Traditional Chinese Medicine Based on Bayesian Method
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Collaborators: Guangzhou University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: haiyin huang
Record Dates: First submitted 2020-08-24; First posted 2020-10-26 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-09

CONDITIONS: Bronchiectasis; Quality of Life; Traditional Chinese Medicine; Sputum; Symptoms; Individuality
Keywords: N-of-1 trials; Drugs, Chinese Herbal; symptoms; individualized treatment; stable bronchiectasis; Bayesian
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, crossover comparisons of individualized herbal decoction with control decoction within individual patients. Each N-of-1 trial has 3 pairs of treatment periods. The duration of each treatment period will be 4 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo is made by dextrin, bitter agent, edible pigment etc and added 5% test drug. The test drug and control drug have no differences in dosage form, appearance, color, specification, label, and so forth.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Individualized Decoction (Experimental): It is the highly individualized treatment of TCM, the modification of Bronchiectasis Stabilization Decoction (Rhizoma Fagopyri Cymosi 30g, Radix Lithospermi 15g, Radix Ophiopogonis 15g, Poria cocos 15g, Radix Astragali 20g, Rhizoma Bletillae 10g, Platycodon grandiflorum 10g, Semen Coicis 30g) based on syndrome differentiation. For subjects with lung and spleen qi deficiency syndrome, the investigators added Radix Codonopsis Pilosulae, Pericarpium Citri Reticulatae, and Atractylodes Macrocephala Koidz. The investigators can adjust the individualized decoction in accordance with the change in the patient's condition throughout the whole study duration.
  The Chinese herbal decoction is taken by one decoction a day and divided into 2 doses, for 3 weeks in each observation period.
  Interventions: Drug: Individualized Decoction; Drug: placebo; Drug: Tested drug minus heat-clearing herbs
- placebo (Placebo Comparator): Placebo is made by dextrin, bitter agent, edible pigment etc. and added 5% test drug. The placebo and test drug have no differences in dosage form, appearance, color, specification, label, and so forth.
  The placebo is taken by one decoction a day and divided into 2 doses, for 3 weeks in each observation period.
  Interventions: Drug: Individualized Decoction; Drug: placebo
- Tested drug minus heat-clearing herbs (Active Comparator): It is the decoction of the Individualized Syndrome Differentiation Decoction (tested drug) minus heat-clearing herbs. For example, heat-clearing herbs such as Scutellaria Baicalensis, Rhizoma Coptidisor Herba Violae will be removed from the Syndrome Differentiation Decoction.
  This control Chinese herbal decoction is taken by one decoction a day and divided into 2 doses, for 3 weeks in each observation period.
  Interventions: Drug: Individualized Decoction; Drug: Tested drug minus heat-clearing herbs

INTERVENTIONS:
Drug: Individualized Decoction — Applied in the Tested Drug Observation Period. It is the highly individualized treatment of TCM, the modification of Bronchiectasis Stabilization Decoction (Rhizoma Fagopyri Cymosi 30g, Radix Lithospermi 15g, Radix Ophiopogonis 15g, Poria cocos 15g, Radix Astragali 20g, Rhizoma Bletillae 10g, Platycodon grandiflorum 10g, Semen Coicis 30g) based on syndrome differentiation. For example, for patients with qi and yin deficiency syndrome, the investigators added Adenophora Root, Radix Glehniae and Radix Rehmanniae Recens etc. For patients with phlegm-heat syndrome, the investigators added Radix Scutellariae and Viola Yedoensis etc. Besides, the herbs in a prescription could be changed according to different symptoms of individual patients.
  Other Names: Syndrome Differentiation Decoction
Drug: placebo — Applied in the placebo Observation Period. Placebo is made by dextrin, bitter agent, edible pigment etc. and added 5% test drug. The test drug and control drug have no differences in dosage form, appearance, color, specification, label, and so forth.
  Arms: Individualized Decoction; placebo
Drug: Tested drug minus heat-clearing herbs — It is the decoction of the Syndrome Differentiation Decoction (tested drug) minus heat-clearing herbs. For example, heat-clearing herbs such as Scutellaria Baicalensis, Rhizoma Coptidisor Herba Violae will be removed from the Syndrome Differentiation Decoction.
  Arms: Individualized Decoction; Tested drug minus heat-clearing herbs

SUMMARY:
The guiding role of parallel randomized controlled trials in clinical practice is limited due to the insufficiency of individual information. Our previous studies showed that Single case randomized controlled trials (referred to as N-of-1 trials) could reflect the individualized characteristics of traditional Chinese medicine (TCM) syndrome differentiation with good feasibility, but the sensitivity was low.

This study aims to compare the efficacy of treatment based on syndrome differentiation with controlled decoctions (placebo, and the method of strengthening the body resistance and removing phlegm) among patients with stable bronchiectasis through a series of N-of-1 trials (single-patient, double-blind, randomized, multiple crossover design), with the 7 point-likert scale of the most concerned symptoms as the main outcome. Hierarchical Bayesian statistical methods and some parameters and variables will be introduced, such as TCM syndrome type, potential residue effect of TCM, etc. The sensitivity and applicability of various mathematical models (Hierarchical Bayesian, paired t-test and Meta-analysis) for N-of-1 trials of TCM will be tested, for the purpose of improving the sensitivity and applicability of N-of-1 trials of TCM both on individual and group levels.

DETAILED DESCRIPTION:
TCM has made great progress in the context of modern science and technology, but compared with the rapid development of modern medicine, the development of TCM has been relatively slow. The randomized controlled trial based on population is incompatible with the characteristics of TCM syndrome differentiation. The lack of reliable efficacy evaluation methods based on evidence-based medicine has hindered the internationalization and development of TCM.

The clinical trial (International clinicaltrials.gov Identifier: NCT03147443) the investigators just finished found that the improved mixed effects model can detect the residual effect of TCM in the N-of-1 trials and improve the sensitivity of group data statistics. However, the sensitivity of this study method is low at the individual statistical level due to the inherent nature of N-of-1 trials, and more cases need to be studied for further improvement. Now that hierarchical Bayesian statistical method has become one of the major statistical methods in a series of N-of-1 trials. Compared with the frequentist statistical methods, the advantages of Bayesian method are as follows: (1) the integration analysis of both individual and group data can be carried out at the same time; (2) it is easy to introduce confounding variables, such as the physique or gene type of different subjects, or different TCM syndrome types (which are helpful to distinguish different TCM syndrome types and the difference of the effects); (3) in addition, there is a special advantage: if a large number of patients have completed similar N-of-1 trials with the variance within an individual patient greater than that between the patients, through "borrowing from strength" , the results of other patients can be used to improve the accuracy of an individual result, that is, to improve the sensitivity of N-of-1 trials, without the need to increase the pairs of N-of-1 trials. At present, this statistic method is rarely used in N-of-1 trials of TCM, so it is worth using for reference in our future research.

The key hypothesis of this study is that: (1) the efficacy of syndrome differentiation will be better than placebo in patients with stable bronchiectasis through N-of-1 trials. (2) the efficacy of syndrome differentiation will be better than the same prescription minus heat-clearing Chinese herbs in patients with stable bronchiectasis through N-of-1 trials. However, at the individual level, with the severity of individual phlegm heat, the efficacy will be different, reflecting the effect of individual treatment based on syndrome differentiation of Chinese medicine. (3) Hierarchical Bayesian statistical model will improve the sensitivity and applicability of N-of-1 trials of TCM both on individual and group levels.

In this study, the investigators will conduct a single center N-of-1 trials in 71 patients with stable bronchiectasis without hemoptysis and respiratory failure. These N-of-1 trials will be randomized, double-blind, crossover comparisons of individualized herbal decoction with control decoction within individual patients. Each N-of-1 trial will have 3 pairs of treatment periods. The duration of each treatment period will be 4 weeks. The investigators will compare: (1) the efficacy of syndrome differentiation (individualized decoction) with placebo, (2) the efficacy of syndrome differentiation (individualized decoction) with the same prescription minus heat-clearing Chinese herbs, in patients with stable bronchiectasis through a series of N-of-1 trials. The primary outcome is patient self-reported symptoms (such as cough, expectoration, shortness of breath, chest pain, and fatigue) scores on a 7 point likert scale. Secondary outcomes are 24-hour sputum volume and the chronic obstructive pulmonary disease (COPD) Assessment Test (CAT) scores. Hierarchical Bayesian statistical methods and some parameters and variables will be introduced, such as TCM syndrome type, potential residue effect of TCM, etc. The sensitivity and applicability of various mathematical models (Hierarchical Bayesian, paired t-test and Meta-analysis) for N-of-1 trials of TCM will be tested, for the purpose of improving the sensitivity and applicability of N-of-1 trials of TCM both on individual and group levels.

ELIGIBILITY:
Inclusion Criteria:

* according to the consensus of domestic experts, combined with the guidelines for the management of adult bronchiectasis published by the European Respiratory Society in 2017;
* male or female, aged 18-70 years;
* being in the stable stage, and no acute exacerbation of bronchiectasis within the past three weeks;
* frequency of acute exacerbation of bronchiectasis ≤3 times every year;
* signed informed consent for participation.

Exclusion Criteria:

* failing to meet the above criteria for diagnosis and inclusion;
* having developed respiratory failure with estimated survival time less than one year;
* having hemoptysis as a comorbidity;
* having complications by active tuberculosis;
* being pregnant or with severe heart, liver, or kidney dysfunctions;
* participating in other pharmacological clinical trials within the past 3 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient Self-Rated Symptom Score (likert scale) | 4 weeks
  Patients rated the severity of the symptoms (such as cough, expectoration, shortness of breath and chest pain) on a 7 point likert scale. Optimize the number of questions to ensure that the most important aspects of the patient's problem are detected (usually four to eight items). Every day each patient scored the severity of these problems on the 7 point Likert scales supplemented by Visual Analogue Scales (VAS). The higher the score, the more severe the symptom.
  The investigators consider an improvement of 0.5 points per question corresponds to a noticeable improvement in the patient's well-being. If there are seven questions, a total change of 3.5 or more points is considered clinically significant. Thus the mean difference of 0.5 points was defined as the "Minimal Clinically Important Difference (MCID)" for the 7 point scales.

SECONDARY OUTCOMES:
24 hours sputum volume | 4 weeks
  The investigators measured the 24h sputum volume at the beginning and the end of each treatment period of the trial. To ensure the accuracy of the measurement, the investigators asked the patients to spit sputum into a collector with scales from 8:00 am to the next 8:00 am. The investigators used the mean value of the sputum volume for 3 consecutive days as the outcome.
COPD Assessment Test (CAT) | 4 weeks
  The CAT had been proven to be effective and reliable in patients with bronchiectasis. CAT questionnaire is composed of 8 items. Each item has a score ranging from 0 to 5, thereby making the total score range from 0 to 40. Score of 0 represents the best quality of life and 40 does the worst. The MCID for the CAT has not been established officially, but it was estimated to be around 2 points.

OTHER OUTCOMES:
Treatment preference for TCM | Through study completion, an average of half a year
  Proportion of patients who prefer to continue TCM treatment after the conclusion of the N-of-1 trial.
Change in of the alanine aminotransferase (ALT), to evaluate the safety of TCM treatment | Baseline and month 6
  Alanine aminotransferase, ALT in U/L.
Change in of the blood urea nitrogen (BUN), to evaluate the safety of TCM treatment | Baseline and month 6
  Blood urea nitrogen, BUN in mmol/L.
Change in of the serum creatinine (Scr), to evaluate the safety of TCM treatment | Baseline and month 6
  Serum creatinine, Scr in μmol/L.

CONTACTS AND LOCATIONS:
Locations (1):
- Yueyang Hospital of Integrated Traditional Chinese and Western Medicine, Shanghai University of Traditional Chinese Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share individual participant data (IPD) with other researchers
Supporting Information: Study Protocol, SAP
Time Frame: The data will become available when the investigators finish the study and last for 5 years.
Access Criteria: available to researchers around the world upon request.

REFERENCES:
- [Result] Huang H, Yang P, Wang J, Wu Y, Zi S, Tang J, Wang Z, Ma Y, Zhang Y. Investigation into the Individualized Treatment of Traditional Chinese Medicine through a Series of N-of-1 Trials. Evid Based Complement Alternat Med. 2018 Feb 7;2018:5813767. doi: 10.1155/2018/5813767. eCollection 2018. PMID 29552084
- [Result] Huang H, Yang P, Xue J, Tang J, Ding L, Ma Y, Wang J, Guyatt GH, Vanniyasingam T, Zhang Y. Evaluating the Individualized Treatment of Traditional Chinese Medicine: A Pilot Study of N-of-1 Trials. Evid Based Complement Alternat Med. 2014;2014:148730. doi: 10.1155/2014/148730. Epub 2014 Nov 11. PMID 25477988
- [Result] Lee BY, Lee S, Lee JS, Song JW, Lee SD, Jang SH, Jung KS, Hwang YI, Oh YM. Validity and Reliability of CAT and Dyspnea-12 in Bronchiectasis and Tuberculous Destroyed Lung. Tuberc Respir Dis (Seoul). 2012 Jun;72(6):467-74. doi: 10.4046/trd.2012.72.6.467. Epub 2012 Jun 29. PMID 23101012
- [Result] Guyatt G，Rennie D. Users'Guides to the Medical Literature: A Manual for Evidence-Based Clinical Practice[M].Chicago: American Medical Association Press，2002:3-11.
- [Result] Dodd JW, Hogg L, Nolan J, Jefford H, Grant A, Lord VM, Falzon C, Garrod R, Lee C, Polkey MI, Jones PW, Man WD, Hopkinson NS. The COPD assessment test (CAT): response to pulmonary rehabilitation. A multicentre, prospective study. Thorax. 2011 May;66(5):425-9. doi: 10.1136/thx.2010.156372. Epub 2011 Mar 12. PMID 21398686
- [Result] Jones PW, Price D, van der Molen T. Role of clinical questionnaires in optimizing everyday care of chronic obstructive pulmonary disease. Int J Chron Obstruct Pulmon Dis. 2011;6:289-96. doi: 10.2147/COPD.S18181. Epub 2011 May 26. PMID 21697993
- [Derived] Lu L, An J, Chen H, Yang P, Xu M, Wu Y, Wang Z, Shen L, Chen X, Huang H. A Series of N-of-1 Trials for Traditional Chinese Medicine Using a Bayesian Method: Study Rationale and Protocol. Evid Based Complement Alternat Med. 2021 Apr 17;2021:9976770. doi: 10.1155/2021/9976770. eCollection 2021. PMID 34122611